CLINICAL TRIAL: NCT01598675
Title: Error Based Learning for Restoring Gait Symmetry Post-Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-1240; R21HD068805 (NIH)
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2016-04

CONDITIONS: Stroke
Keywords: stroke; Gait; walking
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Symmetric Gait. Dual-belted treadmill belts moving at the same belt speeds during training
  Interventions: Other: Same Belt Speeds
- Gait Asymmetry (Experimental): Error Augmentation. Belts of a dual-belted treadmill may move at different belt speeds to amplify spatiotemporal gait asymmetry during training
  Interventions: Other: Different Belt Speeds
- Gait Symmetry (Experimental): Error Minimization. Belts of a dual-belted treadmill may move at different belt speeds to encourage spatiotemporal gait symmetry during training
  Interventions: Other: Different Belt Speeds

INTERVENTIONS:
Other: Same Belt Speeds — 18 sessions of training (3X/week). 20 minutes/session on treadmill; 10 minutes/session overground 70-75%HRmax. Control-Dual-belted treadmill belts respond to encourage symmetric gait
  Arms: Control
Other: Different Belt Speeds — 18 sessions of training (3X/week). 20 minutes/session on treadmill; 10 minutes/session overground 70-75%HRmax. Treadmill belts of dual-belted treadmill respond either to amplify asymmetric gait or encourage symmetric gait.
  Arms: Gait Asymmetry; Gait Symmetry

SUMMARY:
Many of the 780,000 people affected by stroke each year are left with slow, asymmetric walking patterns. The proposed project will evaluate the effectiveness of two competing motor learning approaches to restore symmetric gait for faster, more efficient, and safer walking.

DETAILED DESCRIPTION:
Walking after stroke is characterized by reduced gait speed and the presence of interlimb spatiotemporal asymmetry. These step length and stance time asymmetries can be energy inefficient, challenge balance control, increase the risk of falls and injury, and limit functional mobility. Current rehabilitation to improve gait is based on one of two competing motor learning strategies: minimizing or augmenting symmetry errors during training. Conventional rehabilitation often involves walking on a treadmill while therapists attempt to minimize symmetry errors during training. Although this approach can successfully improve gait speed, it does not produce long-term changes in symmetry. Conversely, augmenting or amplifying symmetry errors has been produced by walking on a split belt treadmill with the belts set at different fixed speeds. While this approach produced an 'after-effect' resulting in step length symmetry for short periods of time, with some evidence of long term learning in people with stroke, it had no influence on stance time asymmetry. The investigators propose that patients need real-time proprioceptive feedback of symmetry errors so that they are actively engaged in the learning process. For this project, the investigators developed and validated a novel, responsive, 'closed loop' control system, using a split-belt instrumented treadmill that continuously adjusts the difference in belt speeds to be proportional to the patient's current asymmetry. Using this system, the investigators can either augment or minimize asymmetry on a step-by-step basis to determine which motor learning strategy produces the largest improvement in overground spatiotemporal symmetry.

ELIGIBILITY:
Inclusion Criteria:

* ability to walk >10 m overground without physical assistance
* overground comfortable gait speed (CGS) < 1.0 m/s (using assistive devices and bracing below the knee as needed)
* able to walk independently on the treadmill at >80% CGS
* exhibits stance time and/or step length asymmetry during CGS

Exclusion Criteria:

* cerebellar lesion
* uncontrolled cardiorespiratory/metabolic disease (cardiac arrhythmia, uncontrolled hypertension or diabetes, orthostatic hypertension, chronic emphysema)or other neurological or orthopedic disorders that may affect gait training
* botulinum toxin to the lower limb in the past 6 months
* a history of balance deficits or unexplained falls not related to the stroke
* uncontrolled seizures
* concurrent physical therapy
* Mini-Mental Status Exam (MMSE) < 24
* communication impairments which could impede understanding of the purpose or procedures of the study or an inability to comply with experimental procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in spatiotemporal gait symmetry after 6 weeks of training | participants will be followed for the duration of their training, expected to be about 6 weeks
  Spatiotemporal gait symmetry is calculated as a ratio of paretic to non-paretic measures after walking over a pressure sensitive mat.

SECONDARY OUTCOMES:
Change from baseline in gait speed after 6 weeks of training | participants will be followed for the duration of their training, expected to be about 6 weeks
  Gait speed is measured in m/sec by having participants walk across a 14' pressure sensitive mat.
Change from baseline in balance after 6 weeks of training | participants will be followed for the duration of their training, expected to be about 6 weeks
  Balance will be assessed using the Berg Balance Scale, 4square step test, and the Functional Gait Assessment
Change from baseline in endurance after 6 weeks of training | participants will be followed for the duration of their training, expected to be about 6 weeks
  Endurance will be measured as the distance walked (in meters) during the 6 Minute Walk Test
Change from baseline in quality of life after 6 weeks of training | participants will be followed for the duration of their training, expected to be about 6 weeks
  Quality of Life will be assessed using the Stroke Impact Scale
Change from baseline in metabolic efficiency after 6 weeks of training | participants will be followed for the duration of their training, expected to be about 6 weeks
  Metabolic efficiency is measured as the metabolic cost of transport (MCOT) using a portable metabolic cart to assess cardiorespiratory gas exchange during the 6 Minute Walk Test.
Change from baseline in community ambulation after 6 weeks of training | participants will be followed for the duration of their training, expected to be about 6 weeks
  Community ambulation is assessed using Step Watch Monitors (SAMs) which will be worn daily for a minimum of 7 days during waking hours.
Change from baseline in gait speed at 1 month follow-up | participants will be followed for one month following the duration of their training (expected to be about 6 weeks) for a total of 10 weeks
  Gait speed is measured in m/sec by having participants walk across a 14' pressure sensitive mat.
Change from baseline in balance at 1 month follow up | participants will be followed for one month following the duration of their training (expected to be about 6 weeks) for a total of 10 weeks
  Balance will be assessed using the Berg Balance Scale, 4square step test, and the Functional Gait Assessment
Change from baseline in endurance at 1 month follow up | participants will be followed for one month following the duration of their training (expected to be about 6 weeks) for a total of 10 weeks
  Endurance will be measured as the distance walked (in meters) during the 6 Minute Walk Test
Change from baseline in quality of life at 1 month follow up | participants will be followed for one month following the duration of their training (expected to be about 6 weeks) for a total of 10 weeks
  Quality of Life will be assessed using the Stroke Impact Scale
Change from baseline in metabolic efficiency at 1 month follow up | participants will be followed for one month following the duration of their training (expected to be about 6 weeks) for a total of 10 weeks
  Metabolic efficiency is measured as the metabolic cost of transport (MCOT) using a portable metabolic cart to assess cardiorespiratory gas exchange during the 6 Minute Walk Test.
Change from baseline in community ambulation at 1 month follow up | participants will be followed for one month following the duration of their training (expected to be about 6 weeks) for a total of 10 weeks
  Community ambulation is assessed using Step Watch Monitors (SAMs) which will be worn daily for a minimum of 7 days during waking hours.
Change from baseline in spatiotemporal gait asymmetry at 1 month follow up | participants will be followed for one month following the duration of their training (expected to be about 6 weeks) for a total of 10 weeks
  Spatiotemporal gait symmetry is calculated as a ratio of paretic to non-paretic measures after walking over a pressure sensitive mat.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Lewek, PT, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Ryan HP, Husted C, Lewek MD. Improving Spatiotemporal Gait Asymmetry Has Limited Functional Benefit for Individuals Poststroke. J Neurol Phys Ther. 2020 Jul;44(3):197-204. doi: 10.1097/NPT.0000000000000321. PMID 32516300